CLINICAL TRIAL: NCT06480383
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy, Safety, and Tolerability of ITI-1284 as an Adjunctive Treatment in Patients With Generalized Anxiety Disorder Who Have an Inadequate Response to Generalized Anxiety Disorder Treatment
Brief Title: Study of ITI-1284 as an Adjunctive Treatment in Patients With Generalized Anxiety Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ITI-1284-301
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ITI-1284 10mg (Experimental)
  Interventions: Drug: ITI-1284 10 mg
- ITI-1284 20mg (Experimental)
  Interventions: Drug: ITI-1284 20 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ITI-1284 10 mg — ITI-1284 10 mg tablet, taken once daily, sublingual administration.
  Arms: ITI-1284 10mg
Drug: ITI-1284 20 mg — ITI-1284 20 mg tablet, taken once daily, sublingual administration.
  Arms: ITI-1284 20mg
Drug: Placebo — Matching placebo tablet, taken once daily, sublingual administration
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study evaluating the efficacy, safety, and tolerability of ITI-1284 compared with placebo as adjunctive therapy to GAD treatment in patients meeting Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-5-TR) criteria for GAD who have an inadequate response to ongoing GAD treatment.

DETAILED DESCRIPTION:
The study will be conducted in 3 periods:

* Screening Period (up to 3 weeks) during which patient eligibility will be assessed and the washout of prohibited medications will occur.
* Double-blind Treatment Period (6 weeks) during which patients will be randomized in a 1:1:1 ratio to receive one of the 3 treatments (ITI-1284 10 mg, ITI-1284 20 mg, or placebo).
* Safety Follow-up Period (1 week) during which all patients will return for a safety follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent before the initiation of any study specific procedures;
2. Male or female patients ≥ 18 years of age;
3. At Screening, meet Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-5-TR) diagnostic criteria for moderate or severe GAD as confirmed by the Investigator or Sponsor-approved rater using the Structured Clinical Interview for DSM-5 Clinical Trials Version (SCID-5-CT), and meets all of the following at Screening and Baseline:

   1. HAM-A Total score of ≥ 22;
   2. HAM-A Items 1 (anxious mood) and 2 (tension) scores ≥ 2;
   3. CGI-S score of ≥ 4;
4. History of inadequate response (< 50% improvement in anxiety symptoms as measured by the modified Antidepressant Treatment Response Questionnaire [ATRQ] for GAD) to at least 1 GAD-approved treatment (ie, one of the following GAD-approved treatments: paroxetine, venlafaxine XR, duloxetine, escitalopram, or buspirone) taken at an adequate dose (at least the minimum GAD-approved dose per package insert) and duration (ie, daily for at least 6 weeks) for the treatment of ongoing GAD symptoms;
5. Currently having an inadequate response to one of the following GAD-approved treatments: paroxetine, venlafaxine XR, duloxetine, escitalopram, or buspirone taken at an adequate dose (at least the minimum GAD-approved dose per package insert) and duration (ie, for at least 6 weeks prior to Screening) and agrees to continue the same dosing regimen for the duration of the study.

NOTE: The current GAD-approved treatment must be different from the GAD treatment identified as the historical failure.

Exclusion Criteria:

1. Within the patient's lifetime, has one of the following confirmed DSM-5-TR psychiatric diagnoses:

   1. Schizophrenia, Schizoaffective Disorder, Schizophreniform Disorder or other psychotic disorder;
   2. Bipolar Disorder;
2. MADRS total score > 18 at Screening or Baseline;
3. In the opinion of the Investigator, the patient has a significant risk for suicidal behavior during his/her participation in the study or

   1. At Screening, the patient scores "yes" on Suicidal Ideation Items 4 or 5 of the C-SSRS within 6 months prior to Screening or, at Baseline, the patient scores "yes" on Suicidal Ideation Items 4 or 5 since the Screening Visit;
   2. At Screening, the patient has had 1 or more suicidal attempts within the 2 years prior to Screening;
   3. At Screening or Baseline MADRS Item 10 score ≥ 5; or
   4. The patient is considered to be an imminent danger to him/herself or others based on the assessment of the Investigator.
4. Lifetime history of failure to respond to > 3 of the approved treatments for GAD (ie, paroxetine, venlafaxine XR, duloxetine, escitalopram, or buspirone) at an adequate dose (ie, at least the minimum dose approved for GAD per package insert) and for an adequate duration (ie, at least 6 weeks).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 705 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Hamilton Anxiety Rating Scale (HAM-A) | Week 6
  The HAM-A Scale is a clinician-rated scale measuring both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). It comprises of 14 items that are rated on a 5-point scale ranging from 0 = not present to 4 = very severe, disabling symptoms. The HAM-A total score ranges from 0 to 56 with a higher score indicating increased severity of anxiety symptoms.

SECONDARY OUTCOMES:
Clinical Global Impression Scale-Severity (CGI-S) | Week 6
  The CGI-S is a clinician-rated scale to assess a patient's overall mental health. The scale ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill patients)

CONTACTS AND LOCATIONS:
Locations (60):
- United States (31):
  - Clinical Site, Chandler, Arizona
  - Clinical Site, Encino, California
  - Clinical Site, Glendale, California
  - Clinical Site, Imperial, California
  - Clinical Site, Lemon Grove, California
  - Clinical Site, Oceanside, California
  - Clinical Site, Orange, California
  - Clinical Site, Redlands, California
  - Clinical Site, San Diego, California
  - Clinical Site, Farmington, Connecticut
  - Clinical Site, Gainesville, Florida
  - Clinical Site, Lauderhill, Florida
  - Clinical Site, Maitland, Florida
  - Clinical Site, Miami, Florida
  - Clinical Site, Miami Springs, Florida
  - Clinical Site, Orlando, Florida
  - Clinical Site, Tampa, Florida
  - Clinical Site, Atlanta, Georgia
  - Clinical Site, Decatur, Georgia
  - Clinical Site, Boston, Massachusetts
  - Clinical Site, Ann Arbor, Michigan
  - Clinical Site, Toms River, New Jersey
  - Clinical Site, Brooklyn, New York
  - Clinical Site, North Canton, Ohio
  - Clinical Site, Oklahoma City, Oklahoma
  - Clinical Site, Allentown, Pennsylvania
  - Clinical Site, Media, Pennsylvania
  - Clinical Site, Austin, Texas
  - Clinical SIte, DeSoto, Texas
  - Clinical Site, Plano, Texas
  - Clinical Site, Bellevue, Washington
- Bulgaria (9):
  - Clinical Site, Blagoevgrad
  - Clinical Site, Burgas
  - Clinical Site, Pleven
  - Clinical Site, Plovdiv
  - Clinical Site, Rousse
  - Clinical Site, Sofia
  - Clinical Site, Targovishte
  - Clinical Site, Varna
  - Clinical Site, Vratsa
- Czechia (3):
  - Clinical Site, Brno
  - Clinical Site, Pilsen
  - Clinical Site, Prague
- Finland (4):
  - Clinical Site, Helsinki
  - Clinical Site, Kuopio
  - Clinical Site, Oulu
  - Clinical Site, Tampere
- Poland (6):
  - Clinical Site, Bialystok
  - Clinical Site, Bydgoszcz
  - Clinical Site, Gorlice
  - Clinical Site, Leszno
  - Clinical Site, Poznan
  - Clinical Site, Torun
- Serbia (7):
  - Clinical Site 2, Belgrade
  - Clinical Site 3, Belgrade
  - Clinical Site 4, Belgrade
  - Clinical Site, Belgrade
  - Clinical Site, Kovin
  - Clinical Site, Kragujevac
  - Clinical Site, Novi Kneževac

IPD SHARING:
Plan to Share IPD: No